CLINICAL TRIAL: NCT02483234
Title: Evaluation of Inflammatory and Structural Joint Damage in Patients With Psoriasis and Psoriatic Arthritis Treated With Secukinumab: A Phase 2, Single Arm, Single Centre Mode of Action Study (Psoriasis-Arthritis & Bone Program, PSARTROS)
Brief Title: Psoriasis-Arthritis & Bone Program
Acronym: PSARTROS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Erlangen-Nürnberg Medical School (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CAIN457F2301T
Record Dates: First submitted 2015-06-24; First posted 2015-06-26 (Estimated); Last update posted 2019-09-27 (Actual); Status verified 2019-09

CONDITIONS: Psoriasis; Psoriatic Arthritis
MeSH Terms: conditions — Psoriasis; Arthritis, Psoriatic | interventions — secukinumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Psoriasis/Psoriatic arthritis (Experimental): Patients with Psoriasis and inflammatory and/or structural lesions and/or erosions in the MRI/HR-qCT scan will be treated with Secukinumab. Patients with psoriatic arthritis will be treated with Secukinumab. Bone changes will be evaluated influenced by IL-17 blockade
  Interventions: Drug: secukinumab

INTERVENTIONS:
Drug: secukinumab

SUMMARY:
Purpose and rationale: To define the role of IL-17 as a mediator of structural bone lesions in psoriasis patients and patients with PsA. Primary Objective is the improvement of the PsAMRIS synovitis score baseline vs. week 24.

Drug tested is Secukinumab 300 mg administered weekly for 4 weeks, then 4 weekly s.c. with a duration total of 24 weeks. Indication for this study is Psoriasis (Pso) and psoriatic arthritis (PsA).

ELIGIBILITY:
Inclusion Criteria:

* Patients eligible for inclusion in this study have to fulfill all of the following criteria:

  * Subjects taking DMARDs (e.g. MTX) are allowed to continue their medication if the dose is stable for at least 4 weeks before baseline and should remain on a stable dose up to Week 24.
  * Subjects who have previously been treated with TNFα inhibitors (investigational or approved) will be allowed entry into study after appropriate wash-out period prior to randomization

PsA patients:

* Diagnosis of PsA classified by CASPAR criteria and with symptoms for at least 6 months with moderate to severe PsA who must have at Baseline ≥3 tender joints out of 78 and ≥3 swollen out of 76 (dactylitis of a digit counts as one joint each)
* Rheumatoid factor and anti-CCP antibodies negative at screening
* Subjects with PsA should have taken NSAIDs for at least 4 weeks prior to randomization with inadequate control of symptoms or at least one dose if stopped due to intolerance to NSAIDs
* Subjects taking corticosteroids must be on a stable dose of ≤10 mg/day prednisone or equivalent for at least 2 weeks before baseline and should remain on a stable dose up to Week 24

Psoriasis patients:

* moderate-to severe psoriasis (PASI > 6)
* no diagnosis of PsA
* inflammatory and/or structural lesions and/or erosions in the MRI/HR-qCT scan

Exclusion Criteria:

* • Chest X-ray or chest MRI with evidence of ongoing infectious or malignant process, obtained within 3 months prior to screening and evaluated by a qualified physician

  * Subjects taking high potency opioid analgesics (e.g. methadone, hydromorphone, morphine)
  * Previous exposure to secukinumab or other biologic drug directly targeting IL-17 or IL-17 receptor
  * Ongoing use of prohibited psoriasis treatments / medications (e.g., topical corticosteroids, UV therapy) at baseline. The following wash out periods need to be observed:

    * Oral or topical retinoids 4 weeks
    * Photochemotherapy (e.g. PUVA) 4 weeks
    * Phototherapy (UVA or UVB) 2 weeks
    * Topical skin treatments (except in face, scalp and genital area during screening, only corticosteroids with mild to moderate potency) 2 weeks
  * Subjects who have ever received biologic immunomodulating agents except for those targeting TNFα or IL-23p40, investigational or approved
  * Previous treatment with any cell-depleting therapies including but not limited to anti-CD20, investigational agents (e.g., CAMPATH, anti-CD4, anti-CD5, anti-CD3, anti-CD19)
  * Women of child-bearing potential, defined as all women physiologically capable of becoming pregnant, unwilling to use effective contraception during the study and for a minimum of 20 weeks after stopping treatment. Effective contraception is defined as either:

    * Barrier method: Condom or Occlusive cap (diaphragm or cervical/vault caps) with spermicide (where available). Spermicides alone are not a barrier method of contraception and should not be used alone

The following methods are considered more effective than the barrier method and are also acceptable:

* Total abstinence: When this is in line with the preferred and usual lifestyle of the subject [Periodic abstinence (e.g. calendar, ovulation, symptothermal, post-ovulation methods) and withdrawal are not acceptable methods of contraception]
* Female sterilization: have had a surgical bilateral oophorectomy (with or without hysterectomy) or tubal ligation at least six weeks before taking study treatment. In case of oophorectomy alone, only when the reproductive status of the woman has been confirmed by follow up hormone level assessment
* Use of established oral, injected or implanted hormonal methods of contraception, intrauterine device (IUD) or intrauterine system (IUS). In case of use of oral contraception women should have been stabile on the same pill for a minimum of 12 weeks before taking study treatment.

  * Active ongoing inflammatory diseases other than PsA that might confound the evaluation of the benefit of secukinumab therapy
  * Underlying metabolic, hematologic, renal, hepatic, pulmonary, neurologic, endocrine, cardiac, infectious or gastrointestinal conditions which in the opinion of the investigator immunocompromises the subject and/or places the subject at unacceptable risk for participation in an immunomodulatory therapy
  * History of clinically significant liver disease or liver injury as indicated by abnormal liver function tests such as SGOT (AST), SGPT (ALT), alkaline phosphatase, or serum bilirubin. The investigator should be guided by the following criteria:
* Any single parameter may not exceed 2 x upper limit of normal (ULN). A single parameter elevated up to and including 2 x ULN should be re-checked once more as soon as possible, and in all cases, at least prior to enrollment/randomization, to rule out lab error
* If the total bilirubin concentration is increased above 2 x ULN, total bilirubin should be differentiated into the direct and indirect reacting bilirubin. In any case, serum bilirubin should not exceed the value of 1.6 mg/dL (27 µmol/L)

  * Screening total WBC count <3,000/µL, or platelets <100,000/µL or neutrophils <1,500/µL or hemoglobin <8.5 g/dL (85g/L)
  * Active systemic infections during the last two weeks (exception: common cold) prior to randomization
  * History of ongoing, chronic or recurrent infectious disease or evidence of tuberculosis infection as defined by either a positive PPD skin test (the size of induration will be measured after 48-72 hours, and a positive result is defined as an induration of ≥ 5mm or according to local practice/guidelines) or a positive QuantiFERON TB-Gold test as indicated in the assessment schedule Table 1: Assessment Schedule (Screening to week 24) . Subjects with a positive test may participate in the study if further work up (according to local practice/guidelines) establishes conclusively that the subject has no evidence of active tuberculosis. If presence of latent tuberculosis is established then treatment according to local country guidelines must have been initiated.
  * Known infection with HIV, hepatitis B or hepatitis C at screening or randomization
  * History of lymphoproliferative disease or any known malignancy or history of malignancy of any organ system within the past 5 years (except for basal cell carcinoma or actinic keratoses that have been treated with no evidence of recurrence in the past 3 months, carcinoma in situ of the cervix or non-invasive malignant colon polyps that have been removed)
  * History or evidence of ongoing alcohol or drug abuse, within the last six months before randomization
  * Plans for administration of live vaccines during the study period or within 6 weeks preceding randomization.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2015-05-31 (Actual); Primary Completion 2018-06-30 (Actual); Study Completion 2018-09-30 (Actual)

PRIMARY OUTCOMES:
The improvement of the PsAMRIS synovitis score | baseline to week 24

CONTACTS AND LOCATIONS:
Locations (1):
- University of Erlangen-Nuremberg, Erlangen, Germany

REFERENCES:
- [Derived] Kampylafka E, Tascilar K, Lerchen V, Linz C, Sokolova M, Zekovic A, Kleyer A, Simon D, Rech J, Sticherling M, Schett G, Hueber AJ. Secukinumab leads to shifts from stage-based towards response-based disease clusters-comparative data from very early and established psoriatic arthritis. Arthritis Res Ther. 2020 Sep 9;22(1):207. doi: 10.1186/s13075-020-02268-y. PMID 32907626
- [Derived] Kampylafka E, Simon D, d'Oliveira I, Linz C, Lerchen V, Englbrecht M, Rech J, Kleyer A, Sticherling M, Schett G, Hueber AJ. Disease interception with interleukin-17 inhibition in high-risk psoriasis patients with subclinical joint inflammation-data from the prospective IVEPSA study. Arthritis Res Ther. 2019 Jul 26;21(1):178. doi: 10.1186/s13075-019-1957-0. PMID 31349876
- [Derived] Kampylafka E, d'Oliveira I, Linz C, Lerchen V, Stemmler F, Simon D, Englbrecht M, Sticherling M, Rech J, Kleyer A, Schett G, Hueber AJ. Resolution of synovitis and arrest of catabolic and anabolic bone changes in patients with psoriatic arthritis by IL-17A blockade with secukinumab: results from the prospective PSARTROS study. Arthritis Res Ther. 2018 Jul 27;20(1):153. doi: 10.1186/s13075-018-1653-5. PMID 30053825